CLINICAL TRIAL: NCT03146156
Title: Lifestyle Intervention in Preparation for Pregnancy (LIPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pennington Biomedical Research Center (Other); The Cleveland Clinic (Other); MetroHealth Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB16-00553; R01HD088061 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-05-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Lifestyle-related Condition; Macrosomia, Fetal
Keywords: obesity; overweight; lifestyle intervention; fetal growth/adiposity; Mediterranean diet
MeSH Terms: conditions — Obesity; Mental Disorders; Fetal Macrosomia; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): Lifestyle coaches will provide personalized instruction on physical activity, dietary data, and behavioral strategies.
  Interventions: Behavioral: Lifestyle Intervention
- Usual Care (No Intervention): The usual care/control groups will be followed by their primary Obstetrical provider. All overweight/obese women will be offered nutrition counseling early in pregnancy by a registered dietician to support GWG within the IOM guidelines.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The lifestyle intervention is healthy eating (Medeterranian diet) and exercise to decrease weight by 5-7% compared to prepregnancy weight.
  Arms: Lifestyle Intervention

SUMMARY:
Studies evaluating lifestyle intervention in obese women during pregnancy have reported limited success in decreasing excessive gestational weight gain, and have failed to achieve the key outcome of breaking the obesity cycle and reducing neonatal adiposity or birth weight. Although some investigators advocate weight loss during pregnancy in obese women, these recommendations were based on extrapolation of retrospective epidemiological data. Of concern, we reported increased small for gestational age babies and decreased lean body mass in neonates of obese women with weight loss or inadequate gestational weight gain. Based on our research, optimal outcomes from lifestyle interventions are likely to be temporal and therefore must be initiated prior to conception to first improve maternal metabolic function, and subsequently, placental/fetal growth. Several large retrospective cohort studies support our hypothesis. For example, women who lost weight between pregnancies had fewer large for gestational age babies in contrast to women who increased interpregnancy weight. In addition, prospective randomized controlled trials have shown that postpartum weight loss is achievable without adverse maternal or neonatal outcomes, these studies include women who breastfed. Based on these observations, we propose a randomized control trial to determine the effect of lifestyle intervention initiated prior to a planned pregnancy on improving neonatal metabolism and adiposity. Our overarching hypothesis is that the maternal pre-pregnancy metabolic condition determines the obesogenic in-utero environment, which affects programming of placental mitochondrial function and metabolic pathways, promoting lipid accumulation and neonatal adiposity. Our rationale is based on the need to establish the most effective time to introduce an intervention that will break the obesity cycle in mothers and their children. Understanding how pregravid metabolic conditioning improves maternal physiology, and cellular and molecular function in pregnancy will provide the empirical data to support the intervention. We have a highly successful record of recruiting women who are planning a pregnancy, obtaining compliance in longitudinal studies, and in long-term follow-up of mothers and their offspring. Lifestyle intervention will be initiated prior to conception to decrease maternal body fat, inflammation, insulin resistance, and ?-cell dysfunction. Our transdisciplinary team has the required expertise in lifestyle interventions management of obesity, and in human physiology that is needed to determine the effects of these interventions on maternal metabolism and fetalplacental growth and function. We will recruit 200 women to pursue the following specific aims:

Specific Aim 1: To investigate the physiological significance of lifestyle intervention in preparation for pregnancy (LIPP) on maternal and neonatal metabolism and adiposity.

Specific Aim 2: To determine the molecular effects whereby lifestyle intervention initiated before pregnancy can improve placental mitochondrial lipid oxidation and accumulation.

DETAILED DESCRIPTION:
Specific Aim 1: To investigate the physiological significance of lifestyle intervention in preparation for pregnancy (LIPP) on maternal and neonatal metabolism and adiposity.

Introduction/Rationale: Our preliminary data demonstrate that supervised lifestyle intervention leads to significant weight loss, improved insulin sensitivity, glucose tolerance and incretin secretion, together with healthier cardiovascular and body composition outcomes in overweight and obese adults. We expect that timing and implementation of the proposed lifestyle intervention will produce similar health benefits in overweight/obese women planning a second pregnancy, and lead to greater insulin sensitivity, reduced insulin secretion, and less inflammation. These improvements will result in the prevention of excess nutrient availability (glucose and lipids) from contributing to excess fetal growth/adiposity. The working hypothesis for this Aim is that in contrast to GWG, the decreased pre-pregnancy insulin sensitivity in obese mothers accounts for the greatest clinical variance in fat accretion in the infant. Although clinically we anticipate a decrease in weight and BMI in the LIPP group, the improvement in insulin sensitivity and metabolic profile are the key physiological measures related to the primary outcome of decreased neonatal adiposity, and not the weight loss per se.

The rationale is that the optimal time to implement lifestyle intervention that effectively improves maternal health at the physiological, cellular and molecular level, and results in optimal adiposity in the baby, is prior to pregnancy. Women who lose weight postpartum, experience a decrease in neonatal birth weight (primarily adipose tissue) in subsequent pregnancy, whereas women who gain weight, experience an increase in neonatal birth weight and adiposity. We hypothesize that maternal pre-pregnancy metabolic condition determines the obesogenic in-utero environment, which in turn affects placental programming of mitochondrial and lipid pathways (Specific Aim 2), and body composition of the baby. An additional rationale is that there is a need to understand how improved pregravid metabolic condition affects maternal physiological and molecular function. We anticipate that obese women who complete the LIPP program will enter pregnancy with improved insulin regulated metabolism and reduced insulin resistance, thus facilitating a lower neonatal birth weight and adiposity. We will recruit mothers who delivered their first baby at MHMC. We recognize that these mothers represent a demographic that has limited access to exercise facilities or family support systems that would facilitate free time for exercise. In order to reduce barriers to participation, we will conduct the exercise sessions in local Community Recreation Centers. The Centers have child care facilities and we will support the cost so participants may bring their babies to the LIPP sessions. To further increase participation and maximize retention, we will provide transportation to and from the Recreation Centers. Support for transportation will be requested from the Cleveland Mt. Sinai Foundation. Lifestyle Intervention Weight Loss Phase: The LIPP program is designed to promote weight loss that is 5-10% of body weight. The 4-month weight loss phase consists of aerobic exercise training with diet and behavioral counseling to induce weight loss as was successfully achieved in prior studies. Initially, supervised exercise will be prescribed at 55-60% of HRmax and gradually increased so that after 1-2 weeks, the subjects are exercising at 75-85% of HRmax (~65-70% VO2max). Supervised exercise will consist of walking/jogging on a treadmill and stationary cycling, 3 days/week, 60 min/session (i.e., 500 kcal/session). The women will wear heart rate (HR) monitors (Polar Electro, Woodbury, NY) during each exercise session so that they have visual feedback of their personalized target heart rate goal. Participants will be advised to reduce caloric intake by ~500 kcal/d in order to support their weight loss goals. The recommended diet will provide ~55% of calories as carbohydrate, 25% as fat, and 20% as protein. Participants will be instructed to consume complex carbohydrates and to avoid simple sugars. Specific caloric needs will be estimated by indirect calorimetry and a sedentary (x1.3) physical activity correction factor. Energy intake will be estimated using the food photo diary app, Meal Snap. Digital photography provides an excellent estimate of energy intake (67). Participants who do not own a smart phone will have one provided through support from the Cleveland Foundation.

Records covering a 72-hour diet period will be shared with the research team for determination of calorie and nutrient intake. Meal Snap has a food database of over 350,000 items. However, some meals will not be in this database, therefore our Lifestyle Coaches will enter all foods eaten into our diet database (NDSR, Minneapolis, MN) to facilitate analysis of calorie, and macro/micro nutrient intake. Subjects will generate photos from before and after the meal in order to estimate the amount of food that was eaten. Data will be obtained at baseline, and at 2-week intervals during the initial 16-week supervised weight loss period.

Lifestyle Intervention - Weight Management/Maintenance: The pre-pregnancy weight management program (phase 2A, 2B and 2C) is designed to facilitate personalized weight loss goals using lifestyle behaviors that include, exercise, diet and behavioral modification, and is based in part on the Look AHEAD trial. The intervention includes a toolbox concept to help meet weight loss goals. The Lifestyle Coaches will provide personalized instruction on physical activity/exercise - 10,000 steps/day, and the participants will use FitBit Flex (Fitbit.com), to track step count and exercise time. During the first phase of weight maintenance (2A) the women will attend 2 supervised group sessions/week. These sessions include structured exercise (e.g., Zumba, jazzercise, stroller walking), review of dietary photo records, where meals have been eaten (home or away; recorded on smart phone app), and behavioral counseling (with their Lifestyle Coach). Participants will be encouraged to eat 1,200-1,500 kcal/d (~55% carbohydrate, 25% fat, 20% protein) if below 113 kg, or 1,500-1,800 kcal/d if >113 kg. Dietary data will be analyzed at 4-week intervals during the weight maintenance period. Importantly, to minimize subject burden and to maximize retention and data acquisition, the Lifestyle Coach will track calorie intake using the participant's photo diary. Behavioral strategies to motivate healthy lifestyle decisions will include: self-monitoring (food, activity, and weight, using FitBit online resources), goal setting (steps/day, weight loss), stimulus control (i.e., social eating, fast food, sitting vs. standing), problem solving (have snacks available, exercise at home), and relapse prevention (i.e., holidays, alcohol, fast food, sweets, problem foods, compulsive eating). After 4 months and the desired weight loss, subjects move to Phase 2B. During this phase subjects maintain an exercise goal of 10,000 steps/day, but will be required to attend only 1 supervised session/week. If a subject fails to maintain weight loss, defined as weight gain of 3% of current body weight, participants will return to Phase 2A for more supervised weight management. Alternatively, if weight loss is maintained after 3 months, subjects will progress to Phase 2C until the subsequent pregnancy. Phase 2C consists of no supervised exercise sessions. However, the subject and Lifestyle Coach will converse weekly by phone to review progress, including Fitbit exercise data and diet. Data suggest that weight management programs delivered by phone are comparable to clinically delivered programs. During the calls participants will be counseled to continue to exercise at the intensity and duration prescribed during Phase 2B. They will be provided with language-specific food and exercise log books. These will be used to guide calorie intake and will provide another record of compliance. Participants randomized to the Control group will receive information on post-pregnancy diet/weight loss from the CRU nutritionist as distinct from the LIPP nutritionist (HB) to decrease cross contamination between groups. Weight Management during Pregnancy: All LIPP and usual care/control groups will be followed by their primary Obstetrical provider. The OB/GYN department at MHMC has recently revised its clinical guidelines for the management of the overweight/obese women based on the December 2015 ACOG practice bulletin (2). All overweight/obese women will be offered nutrition counseling early in pregnancy by a registered dietician from the MHMC Nutrition Department with follow-up visits as needed to support GWG within the IOM guidelines. Nutritional therapy will consider maternal pregravid BMI, ethnic, cultural and social factors in individualizing healthy eating. The electronic health record (EPIC) includes a graphic GWG nomogram and so GWG will be monitored at each visit. All subjects will be encouraged to increase physical activity for at least 30 minutes/day (primarily walking). Clinical management such as, ultrasounds to estimate fetal growth, and fetal surveillance will be based on the ACOG recommendations. The Lifestyle Coach will continue to follow-up only with the LIPP subjects as described in the maintenance phase of the research design.

Metabolic Evaluations: Metabolic evaluations will be performed at baseline (3 months ? 2 weeks) postpartum. Follow-up evaluations will be performed after 4 (+/-2 weeks) and 12 months (+/-2 weeks), and then every 6 months (+/-2 weeks) prior to pregnancy up to a maximum of 24 months. Once a subject has pregnancy dating and viability confirmed by ultrasound, metabolic evaluations will continue at 12-16 and 32-36 weeks of gestation.

Maternal Body Composition: Anthropometry measurements will include height, weight, and hip and waist circumferences. Total body fat will be measured by whole body plethysmography (Bod Pod; Cosmed, Rome, Italy). We will use a hydration constant of 76% for fat free mass during late pregnancy.

Resting Energy Expenditure: Resting Metabolic Rate (RMR) will be determined after an overnight fast using the Cosmed OMNIA metabolic cart (Cosmed, Rome Italy) with a canopy system. We will control for diet by providing a standardized energy balanced meal the evening prior to the test from the CRU. Participants will relax in a quiet low-light metabolic room for 30 min prior to obtaining a 30 min measure of exhaled breath. Oxidative and non-oxidative glucose metabolism will be estimated and urine samples will be obtained before and after the measure in order to calculate non-protein RQ (NPRQ). These data will be used in conjunction with Specific Aim 2, and will be correlated with change in mitochondrial function during pregnancy.

Exercise Capacity: An incremental graded treadmill test will be performed at baseline, 4, and 6 month time points in both groups. Oxygen consumption (Jaeger OxyCon Pro/Delta System, Hoechberg, Germany), heart rate, and ratings of perceived exertion will be performed as previously described.

Insulin Sensitivity and ?-Cell Function: A 75 g oral glucose tolerance test (OGTT) will be used to assess postprandial glycemia, and insulin sensitivity and secretion. After an overnight fast, blood samples will be drawn at 10 min intervals for the first 60 min, and at 20 min intervals thereafter. C-peptide data will be analyzed using a combined model approach to provide pre-hepatic insulin secretion rates, insulin sensitivity, disposition index, and relate insulin and Cpeptide kinetics (73). Plasma glucose will be measured using the glucose oxidase method (YSI; Yellow Springs, OH).

Insulin will be assayed by RIA (Millipore, Billerica, MA). Diagnosis of GDM will be made using criteria recommended by the ACOG (74).

Enteroinsular Axis Responses: Plasma samples (with appropriate additives) will be obtained to measure incretin hormones (glucagon-like peptide-1 (GLP-1), and glucose-dependent insulinotropic polypeptide (GIP), and satietyrelated gut peptides (cholecystokinin (CCK), and peptide YY (PYY). Measurements will be made under static (fasting) and dynamic (glucose-stimulated) conditions (10 min intervals up to 1 hour).

Metabolic and Inflammatory Biomarkers: Fasting blood samples will be obtained to measure CBC, TSH, HbA1c, lipid panel, and total free fatty acids (FFA). Adipocytokines (adiponectin, leptin interleukin-6, interleukin- 8, TNF-? and hsCRP) will be measured using ELISA (R&D Systems, Minneapolis, MN). All samples from each subject will be stored at -80oC and run in the same assay at completion to decrease variability.

Quality of Life Questionnaire: The SF-36 health survey will be used at baseline, 4 and 12 months, and then at 6 month intervals until pregnancy to assess the subject's health-related quality of life. These data will provide a generic measure of physical and mental health through assessment of physical functioning, bodily pain, limitations due to physical, personal, or emotional problems and well-being, energy/fatigue, and general health perceptions. During pregnancy the questionnaire will be administered at 12-16 and 32-36 weeks.

Measuring Fat Mass in the Infant: We have extensive experience in estimating body composition in neonates, and were one of the first centers to procure a Pea Pod (pediatric air densitometry), which is housed in the CRU next to Labor & Delivery and the postpartum unit.

Insulin Resistance at Birth: At birth we will obtain umbilical cord blood for insulin and glucose to estimate insulin resistance using HOMA. Full lipid profile, CRP, and the adipokines IL-6 and leptin (an excellent marker of neonatal fat mass) will be measured in cord blood as described above.

Anticipated Results, Challenges, and Alternative Approaches:

The primary outcome measure of this proposal is lower neonatal adiposity at birth in the LIPP group relative to: 1) the Control group and 2) with the subject's firstborn. As secondary outcomes we anticipate that prior to a subsequent pregnancy, LIPP will produce significant improvement (absolute and percent changes) in maternal weight and body composition, and more importantly improved insulin sensitivity, beta-cell function, incretin response to glucose, lipid and inflammatory biomarkers, compared to the Control group. We also expect reduced insulin resistance, cord lipids and inflammatory profiles in babies born to LIPP compared to Controls.

Recruitment is a well-recognized problem for the successful implementation and completion of lifestyle intervention trials. However, given the novel strategy for recruitment detailed above, our unique access to the patient population, and our extensive experience in metabolic research in pregnancy, we do not anticipate recruitment to present an insurmountable challenge. We will recruit 200 subjects in the first 4 years and complete all mother/baby evaluations according to the proposed timeline. If necessary we will recruit subjects from Cleveland Clinic and University Hospitals, both affiliated with Case Western Reserve University (CWRU). Retention strategies include free transportation to the exercise sessions, free childcare service during the lifestyle sessions and consults with the Lifestyle Coach, cell phone apps to reduce subject burden with data entry, regular telephone contacts, and financial incentives, including an infant car seat at delivery.

Our team has had outstanding success in retaining pregnant women in our previous metabolic research and lifestyle intervention studies in overweight and obese populations (48,64). In the current proposal, additional strategies are also in place to maximize retention and minimize dropout. These include phone calls and emails from the Lifestyle Coach to review and reinforce problem solving and self-monitoring skills as described for participants in the Diabetes Prevention Program. We will also establish a buddy system where each participant becomes a buddy to another participant, the two buddies may prepare meals together, exercise together, share problems, etc. The buddy system fosters the sense that staying in the study is important not just for the individual's health but also for the buddy's as well. If subjects in the LIPP program do not meet their target weight loss goal, we will implement a meal replacement strategy using the resources of the CRU/CTSC metabolic kitchen, with attention to the caloric and nutrient needs of the mother depending on breast feeding. Not all participants will conceive. Since the primary outcome is neonatal adiposity, subjects who do not become pregnant will not be included in the primary analysis but will be included in secondary analyses relating to pregravid metabolic improvement. By recruiting women with a previous pregnancy the risk of infertility is significantly reduced. We anticipate that approximately 20% of women will experience a spontaneous abortion, but they will be allowed to continue and resume their previous participation in either the LIPP or Control group. We anticipate that approximately 25% of subjects will drop out before becoming pregnant, and another 15% may drop out during pregnancy. We will enroll 100 subjects in each arm to account for the unlikely event of 40% dropout. Adopting an even more stringent strategy, we report statistical power is available for as low as 50 subjects per group as a worst-case scenario. If retention lags behind projections we will recruit additional subjects at MHMC and CWRU affiliated hospitals. The CRU staff will assist in collecting cord blood and placenta at delivery and performing the Pea Pod body measures. If there is a Pea Pod equipment malfunction we will estimate body composition using neonatal anthropometrics.

Although LIPP subjects will be encouraged to delay a second pregnancy until they are in the maintenance phase of the program, we will exclude LIPP subjects only if they conceive during the first 4 month weight loss phase. For the Control subjects, exclusion will occur if a subject becomes pregnant before the 3 month postpartum CRU randomization visit. Use of birth control in this phase is an inclusion criterion. Not all LIPP subjects will conceive at similar times after the 4 month weight loss intervention. We will not adjust for the time between pregnancies between the LIPP and Control subjects. We will use the LIPP and control subject's metabolic status (body composition, insulin sensitivity and response, etc.) at the last metabolic evaluation in the CRU before becoming pregnant as their pregravid or baseline status for the subsequent pregnancy. Because this is a pregnancy study only women with be recruited. However, we will assess the effect of LIPP on males and female offspring, together and independently, based on sex.

Statistical Approach:

The primary analyses of Specific Aim 1a will be intent-to-treat comparisons of the LIPP and Control groups in regard to changes in maternal insulin sensitivity, BMI, and fat mass. The comparisons will be performed first with two-sample t-tests at p=0.05. Should any imbalance of confounding factors in the groups be recognized, linear regression models that include significant differences (e.g. GDM) will be used to perform covariate adjustments. Based on our 1 year postpartum follow-up studies (62,63), we will have 90% power to detect an absolute or covariate-adjusted improvement in insulin sensitivity of 30% and an 80% power to detect an improvement as small as 25% in the LIPP vs. Control group. Corresponding 95% confidence intervals (95% CI) for the absolute or covariate-adjusted differences or percent improvements in insulin sensitivity between groups will be reported. We estimate the standard deviation (SD) of change in BMI from randomization until subsequent pregnancy to be 5.1 kg/m2. We will have 90% power to detect an absolute or covariate-adjusted difference in BMI of 2.6 kg/m2 and 80% power to detect a difference of 2.26 kg/m2 and 90% power to detect an absolute or covariate-adjusted difference in fat mass of 5.9 kg and 80% power to detect a difference of 5.1 kg between groups prior to the second pregnancy. The primary analysis for Specific Aim 1b is an intent-to-treat comparison of LIPP versus Control neonates with respect to fat mass at birth. The comparison will be performed using a two-sample t-test at p=0.05. Linear regression will be performed, which will include weight (body composition measures) of the subject's first child as a covariate. Should any imbalance of confounding factors (for example gestational age) in the groups be recognized, linear regression models will be used to perform a covariate adjustment. Based on our preliminary data, we estimate the SD of neonatal fat mass between the LIPP and Control groups to be no more than 225g. With at least 50 women in each group, (assuming a 50% dropout), the t-test or linear regression will have 90% power to detect an absolute or covariate-adjusted difference of 146 g fat mass between groups. We have 80% power to detect an absolute or covariate-adjusted difference as small as 126 g fat mass between groups. Corresponding 95% CI for the absolute or covariate-adjusted difference in neonatal fat mass between groups will be reported. For secondary analyses, we will be using the same statistical approach. Based on our preliminary data, we estimate the SD of birth weight to be 700 g; with 50 neonates in each group we will have 90% power to detect an absolute or covariate-adjusted difference of 455 g in birth weight and 80% power to detect a 393 g difference between groups. Additional secondary analyses will include umbilical cord cytokines. Comparisons will be performed using a two-sample t-test at a significance level of p=0.05; however, Mann- Whitney U tests or log transformations will be employed if data are not normally distributed. Linear regression models, including confounding factors, will be used to perform covariate adjustments. Based on our published data (80), we estimate the standard deviations of umbilical cord IL-6 and CRP to be 3.4 pg/ml and 7,900 ng/ml, respectively. With 50 women in each group, we will have 90% power to detect an improvement in IL-6 and CRP levels of 50% and 42%, and 80% power to detect an improvement of 42% and 36%, respectively.

Specific Aim 2: To determine the molecular effects whereby lifestyle intervention initiated before pregnancy can improve placental mitochondrial lipid oxidation and accumulation.

Introduction/Rationale: Our data suggest that in obese women, a mitochondrial defect in placental tissue is present early in pregnancy, inhibiting the placental capacity for fatty acid oxidation and shunting fatty acids to esterification pathways and lipid accumulation, potentially leading to increased nutrient availability to the fetus and higher adiposity at term. Our group has shown that other mitochondrial processes, such as cholesterol transport and steroidogenesis are impaired in placentas of obese, insulin resistant women at term. Placental mitochondrial content (assessed by mtDNA and citrate synthase activity) is not affected by maternal obesity and insulin resistance at term, suggesting that the observed defects in function are due to changes in mitochondrial activity, rather than number. Previous dietary interventions initiated during pregnancy were unable to alter placental ?-oxidation or fetal fat deposition, potentially because the intervention was begun after placental mitochondrial function was impaired. We anticipate that LIPP will improve placental mitochondrial fatty acid oxidation, which will be measurable at term and associated with lower fatty acid esterification and accumulation, and neonatal fat mass. The hypothesis is that the decreased insulin sensitivity and increased inflammatory environment in obese mothers impairs mitochondrial ?-oxidation in the developing placenta. It is the changes in placental metabolism beginning early in pregnancy that lead to altered nutrient delivery and increased fetal fat deposition. Our rationale is based on the need to understand how changes in placental lipid metabolism mediate the effects of improved pregravid metabolism on neonatal adiposity. We expect that placentas of obese women in the LIPP program will show improved fatty acid oxidation and decreased lipid esterification and accumulation at term. Furthermore, we expect that these changes will correlate with lower maternal inflammation and insulin resistance in early pregnancy and lower neonatal adiposity at term.

Anticipated Results and Endpoints: We anticipate that compared to the Control group, placentas of women in LIPP will have: 1) increased ?-oxidation, 2) decreased fatty acid esterification, 3) lower lipid content, 4) increased activity of mitochondrial CPT1B, the rate-limiting enzyme in ?-oxidation, and higher phosphor ACC, which, when phosphorylated, produces less malonyl CoA, the main inhibitory regulator of CPT1B, and 5) no difference in mitochondrial content (as measured by mtDNA and citrate synthase activity). We also anticipate that mitochondrial ?-oxidation and CPT1B activity will negatively correlate with early pregnancy maternal serum inflammatory cytokine markers and insulin resistance and neonatal adiposity.

Experimental Design: We will accomplish the objectives of Specific Aim 2 by measuring changes in placental mitochondrial enzyme activity and lipid metabolism in women enrolled in the Control or LIPP groups described in Specific Aim 1. Placental tissue will be collected at delivery from all study participants and embedded in paraffin, or snap frozen in liquid nitrogen, and stored at -80oC for molecular analysis. In a subset of women delivering by scheduled Cesarean delivery (we estimate ~30% of our participants or N=15-18/group), we will also collect fresh placental tissue for lipid metabolism activity assays.

Placental lipid metabolism: These assays are well established in the O'Tierney-Ginn lab. Mitochondrial fatty acid oxidation (FAO) and esterification into total lipid assays will be performed in placental explants as described previously, with some modifications. Freshly isolated placental explants will be incubated in the presence of 100 ?M cold palmitate and 3H-palmitate (Moravek Radiochemicals) for 18 hrs. At the end of the incubation period, media will be collected to quantify the FAO rate by detection of 3H2O using the vapor phase equilibration method of Hughes. Esterificationinto total lipids will be determined by homogenizing the treated explants in HPLC-grade acetone and incubating with agitation at room temperature overnight. An aliquot of the acetone-extract lipid suspension will be used to determine the radioactive content by liquid scintillation counting. Oxidation and esterification rates will be defined as nmol palmitate/mg tissue/hr.

Assessment of placental mitochondria: Mitochondria will be isolated from frozen placental tissue as previously described. Markers of lipid oxidation (CPT1B) and synthesis/esterification (phospho-ACC) activity will be measured using commercially available kits (Cell Signaling, Abcam) in isolated mitochondria from all samples. Markers of mitochondrial content (mtDNA and citrate synthase activity) will be measured in whole placental tissue in all samples as previously described.

Placental Lipid Accumulation: Total placental lipid content will be measured using the Folch method.

Anticipated Challenges and Alternatives: 1) We will use only placentas delivered by scheduled cesarean delivery for in vitro oxidation and esterification assays, to avoid changes pertinent to labor. At our hospital, the rate of cesarean for obese women is ~40%. Our conservative estimate of 40-50% drop-out followed by 30% of subjects delivering by cesarean, results in N=15-18/group. Based on our preliminary data, this will leave us adequately powered to detect differences in placental lipid metabolism due to LIPP. We will collect placental samples from all study participants for mitochondrial enzyme activity assays, providing us with an additional assessment of metabolic activity in a larger number of participants. 2) Placental mitochondrial fatty acid oxidation capacity may be affected by mitochondrial number, oxidative phosphorylation activity, and energetic efficiency (coupling). Assessment of mitochondrial oxidative phosphorylation capacity or energetic efficiency requires freshly isolated mitochondria and/or living cells which, for our proposal, would be overly ambitious and costly considering the unpredictable nature of delivery and the large number of participants. Alternatively, we will measure markers of mitochondrial content and key enzymes in mitochondrial lipid metabolism in all placental samples to assess some potential mechanisms underlying changes in placental fatty acid oxidation. Additionally, frozen samples collected from all placentas can be used to measure enzymes involved in electron transport (e.g., ATP synthase) as a marker of mitochondrial oxidative phosphorylation.

Statistical Analysis: The primary goal of Aim 2 is to determine the effect of lifestyle intervention prior to pregnancy on placental mitochondrial fatty acid oxidation at term. We hypothesize that placental ?-oxidation will be higher in the LIPP group. We will conduct an intent-to-treat analysis using two sample t-test or non-parametric Wilcoxon rank-sum test to assess differences between groups. Regression analysis will be used to assess the association of placental ?-oxidation and enzyme activity with maternal inflammatory cytokine levels and insulin resistance in early pregnancy, along with neonatal fat mass with adjustment for gestational age and gender. Descriptive statistics, such as mean, median and range will be calculated for all variables. Power and sample size analysis based on our preliminary mitochondrial ?-oxidation data in obese women (38?14 nmol/mg/hr) showed that a sample size of N=18/group achieves 80% power to detect a difference of 25% between groups using a two-sample t-test with a significance level of 0.05.

ELIGIBILITY:
Inclusion criteria:

All subjects will have had by the time of randomization at 3 months postpartum:

1. Planning another pregnancy within the next 24 months
2. Planning to deliver at Tufts medical center during their next pregnancy
3. A previous full-term singleton pregnancy (gestational age > 37 weeks)
4. 18 to 40 years of age at the time of enrollment into the study
5. Vaginal or cesarean delivery
6. Normal glucose tolerance or gestational diabetes (GDM), but without evidence of postpartum diabetes as defined by a 75 g 2-hr oral glucose tolerance test (OGTT)
7. Normal blood pressure or mild preeclampsia but normal postpartum blood pressure
8. Bottle or breast feeding
9. Normal thyroid function (determined by TSH concentration in blood), normal cell blood count and normal kidney and liver functions. Lipid profile with triglyceride levels not higher than 400 mg/dl (fasting) and LDL levels less than 180 mg/dL
10. No clinical signs or symptoms of cardiovascular disease or any other disease or condition that may contraindicate participation in exercise training (i.e. COPD, severe asthma, orthopedic abnormalities)
11. Using contraception

Exclusion criteria:

1. Pre or post-delivery diabetes
2. Post-delivery hypertension requiring medication
3. asthma requiring more than occasional use of a sympathomimetic inhaler, but not chronic inhaled steroids
4. Inflammatory bowel disease
5. Need for assisted reproductive technologies to become pregnant
6. Medical or obstetrical contraindication to the defined exercise program or diet
7. Tobacco, excessive alcohol use (greater than 2 drinks/day) or illicit drug use
8. Eating disorders such as bulimia
9. Gastric surgery to lose weight including banding or bypass procedures
10. Any psychological or psychiatric condition which may impair participation in the lifestyle intervention program
11. Multiple pregnancy
12. HIV, or hepatitis B or C
13. If a LIPP subject becomes pregnant prior to 16 weeks after randomization before the weight- loss phase for the lifestyle intervention is completed or a control subject becomes pregnant before the 3 month postpartum randomization, i.e. no baseline measurement.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We will recruit a total of 200 overweight/obese subjects (defined as pregravid BMI 25-35 kg/m2) at the time of their first pregnancy, hereafter defined as obese for the purposes of the proposal) determined by review of the electronic medical record (EMR) after delivery of their first child.
Enrollment: 99 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Neonatal adiposity comparison between intervention and usual care group | 48 to 72 hours after delivery
  Neonatal anthropometry and air densitometry (pea pod)

SECONDARY OUTCOMES:
Maternal metabolic status | from baseline to 6 month post-partum and then during pregnancy at 12 to 16 weeks gestation and 34 to 36 weeks gestation.
  body composition, insulin sensitivity and insulin response

CONTACTS AND LOCATIONS:
Overall Officials: Li Yin Cheok, MA, Study Director — Tufts Medical Center
Locations (4):
- United States (4):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be available in a de-identified manner by contacting the Principal Investigator, after the results have been published.
Time Frame: The results of the study will be available in a de-identified manner by contacting the Principal Investigator, after the results have been published.
Access Criteria: The results of the study will be available in a de-identified manner by contacting the Principal Investigator, after the results have been published.

REFERENCES:
- [Background] Magkos F, Fraterrigo G, Yoshino J, Luecking C, Kirbach K, Kelly SC, de las Fuentes L, He S, Okunade AL, Patterson BW, Klein S. Effects of Moderate and Subsequent Progressive Weight Loss on Metabolic Function and Adipose Tissue Biology in Humans with Obesity. Cell Metab. 2016 Apr 12;23(4):591-601. doi: 10.1016/j.cmet.2016.02.005. Epub 2016 Feb 22. PMID 26916363
- [Background] ACOG Practice Bulletin No 156: Obesity in Pregnancy. Obstet Gynecol. 2015 Dec;126(6):e112-e126. doi: 10.1097/AOG.0000000000001211. No abstract available. PMID 26595582
- [Background] Finer LB, Zolna MR. Declines in Unintended Pregnancy in the United States, 2008-2011. N Engl J Med. 2016 Mar 3;374(9):843-52. doi: 10.1056/NEJMsa1506575. PMID 26962904
- [Background] Catalano PM. Increasing maternal obesity and weight gain during pregnancy: the obstetric problems of plentitude. Obstet Gynecol. 2007 Oct;110(4):743-4. doi: 10.1097/01.AOG.0000284990.84982.ba. No abstract available. PMID 17906003
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Ananth CV, Wen SW. Trends in fetal growth among singleton gestations in the United States and Canada, 1985 through 1998. Semin Perinatol. 2002 Aug;26(4):260-7. doi: 10.1053/sper.2002.34772. PMID 12211616
- [Background] Surkan PJ, Hsieh CC, Johansson AL, Dickman PW, Cnattingius S. Reasons for increasing trends in large for gestational age births. Obstet Gynecol. 2004 Oct;104(4):720-6. doi: 10.1097/01.AOG.0000141442.59573.cd. PMID 15458892
- [Background] Catalano PM. Management of obesity in pregnancy. Obstet Gynecol. 2007 Feb;109(2 Pt 1):419-33. doi: 10.1097/01.AOG.0000253311.44696.85. PMID 17267845
- [Background] Donahue SMA, Kleinman KP, Gillman MW, Oken E. Trends in birth weight and gestational length among singleton term births in the United States: 1990-2005. Obstet Gynecol. 2010 Feb;115(2 Pt 1):357-364. doi: 10.1097/AOG.0b013e3181cbd5f5. PMID 20093911
- [Background] Gibson KS, Waters TP, Gunzler DD, Catalano PM. A retrospective cohort study of factors relating to the longitudinal change in birth weight. BMC Pregnancy Childbirth. 2015 Dec 22;15:344. doi: 10.1186/s12884-015-0777-8. PMID 26693917
- [Background] Rasmussen KM, Abrams B, Bodnar LM, Butte NF, Catalano PM, Maria Siega-Riz A. Recommendations for weight gain during pregnancy in the context of the obesity epidemic. Obstet Gynecol. 2010 Nov;116(5):1191-5. doi: 10.1097/AOG.0b013e3181f60da7. PMID 20966705
- [Background] Whitaker RC. Predicting preschooler obesity at birth: the role of maternal obesity in early pregnancy. Pediatrics. 2004 Jul;114(1):e29-36. doi: 10.1542/peds.114.1.e29. PMID 15231970
- [Background] Boney CM, Verma A, Tucker R, Vohr BR. Metabolic syndrome in childhood: association with birth weight, maternal obesity, and gestational diabetes mellitus. Pediatrics. 2005 Mar;115(3):e290-6. doi: 10.1542/peds.2004-1808. PMID 15741354
- [Background] Catalano PM, Farrell K, Thomas A, Huston-Presley L, Mencin P, de Mouzon SH, Amini SB. Perinatal risk factors for childhood obesity and metabolic dysregulation. Am J Clin Nutr. 2009 Nov;90(5):1303-13. doi: 10.3945/ajcn.2008.27416. Epub 2009 Sep 16. PMID 19759171
- [Background] Philipps LH, Santhakumaran S, Gale C, Prior E, Logan KM, Hyde MJ, Modi N. The diabetic pregnancy and offspring BMI in childhood: a systematic review and meta-analysis. Diabetologia. 2011 Aug;54(8):1957-66. doi: 10.1007/s00125-011-2180-y. Epub 2011 May 31. PMID 21626451
- [Background] Walsh JM, McGowan CA, Mahony R, Foley ME, McAuliffe FM. Low glycaemic index diet in pregnancy to prevent macrosomia (ROLO study): randomised control trial. BMJ. 2012 Aug 30;345:e5605. doi: 10.1136/bmj.e5605. PMID 22936795
- [Background] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411
- [Background] Dodd JM, Turnbull D, McPhee AJ, Deussen AR, Grivell RM, Yelland LN, Crowther CA, Wittert G, Owens JA, Robinson JS; LIMIT Randomised Trial Group. Antenatal lifestyle advice for women who are overweight or obese: LIMIT randomised trial. BMJ. 2014 Feb 10;348:g1285. doi: 10.1136/bmj.g1285. PMID 24513442
- [Background] Phelan S, Phipps MG, Abrams B, Darroch F, Grantham K, Schaffner A, Wing RR. Does behavioral intervention in pregnancy reduce postpartum weight retention? Twelve-month outcomes of the Fit for Delivery randomized trial. Am J Clin Nutr. 2014 Feb;99(2):302-11. doi: 10.3945/ajcn.113.070151. Epub 2013 Nov 27. PMID 24284438
- [Background] Renault KM, Norgaard K, Nilas L, Carlsen EM, Cortes D, Pryds O, Secher NJ. The Treatment of Obese Pregnant Women (TOP) study: a randomized controlled trial of the effect of physical activity intervention assessed by pedometer with or without dietary intervention in obese pregnant women. Am J Obstet Gynecol. 2014 Feb;210(2):134.e1-9. doi: 10.1016/j.ajog.2013.09.029. Epub 2013 Sep 20. PMID 24060449
- [Background] Poston L, Bell R, Croker H, Flynn AC, Godfrey KM, Goff L, Hayes L, Khazaezadeh N, Nelson SM, Oteng-Ntim E, Pasupathy D, Patel N, Robson SC, Sandall J, Sanders TA, Sattar N, Seed PT, Wardle J, Whitworth MK, Briley AL; UPBEAT Trial Consortium. Effect of a behavioural intervention in obese pregnant women (the UPBEAT study): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):767-77. doi: 10.1016/S2213-8587(15)00227-2. Epub 2015 Jul 9. PMID 26165396
- [Background] Sagedal LR, Overby NC, Bere E, Torstveit MK, Lohne-Seiler H, Smastuen M, Hillesund ER, Henriksen T, Vistad I. Lifestyle intervention to limit gestational weight gain: the Norwegian Fit for Delivery randomised controlled trial. BJOG. 2017 Jan;124(1):97-109. doi: 10.1111/1471-0528.13862. Epub 2016 Jan 14. PMID 26768233
- [Background] Dodd JM, Grivell RM, Crowther CA, Robinson JS. Antenatal interventions for overweight or obese pregnant women: a systematic review of randomised trials. BJOG. 2010 Oct;117(11):1316-26. doi: 10.1111/j.1471-0528.2010.02540.x. PMID 20353459
- [Background] Tanentsapf I, Heitmann BL, Adegboye AR. Systematic review of clinical trials on dietary interventions to prevent excessive weight gain during pregnancy among normal weight, overweight and obese women. BMC Pregnancy Childbirth. 2011 Oct 26;11:81. doi: 10.1186/1471-2393-11-81. PMID 22029725
- [Background] Quinlivan JA, Julania S, Lam L. Antenatal dietary interventions in obese pregnant women to restrict gestational weight gain to Institute of Medicine recommendations: a meta-analysis. Obstet Gynecol. 2011 Dec;118(6):1395-1401. doi: 10.1097/AOG.0b013e3182396bc6. PMID 22105270
- [Background] Thangaratinam S, Rogozinska E, Jolly K, Glinkowski S, Roseboom T, Tomlinson JW, Kunz R, Mol BW, Coomarasamy A, Khan KS. Effects of interventions in pregnancy on maternal weight and obstetric outcomes: meta-analysis of randomised evidence. BMJ. 2012 May 16;344:e2088. doi: 10.1136/bmj.e2088. PMID 22596383
- [Background] Thangaratinam S, Jolly K. Obesity in pregnancy: a review of reviews on the effectiveness of interventions. BJOG. 2010 Oct;117(11):1309-12. doi: 10.1111/j.1471-0528.2010.02670.x. No abstract available. PMID 20862792
- [Background] Kiel DW, Dodson EA, Artal R, Boehmer TK, Leet TL. Gestational weight gain and pregnancy outcomes in obese women: how much is enough? Obstet Gynecol. 2007 Oct;110(4):752-8. doi: 10.1097/01.AOG.0000278819.17190.87. PMID 17906005
- [Background] Oken E, Kleinman KP, Belfort MB, Hammitt JK, Gillman MW. Associations of gestational weight gain with short- and longer-term maternal and child health outcomes. Am J Epidemiol. 2009 Jul 15;170(2):173-80. doi: 10.1093/aje/kwp101. Epub 2009 May 13. PMID 19439579
- [Background] Bodnar LM, Siega-Riz AM, Simhan HN, Himes KP, Abrams B. Severe obesity, gestational weight gain, and adverse birth outcomes. Am J Clin Nutr. 2010 Jun;91(6):1642-8. doi: 10.3945/ajcn.2009.29008. Epub 2010 Mar 31. PMID 20357043
- [Background] Catalano PM, Mele L, Landon MB, Ramin SM, Reddy UM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Saade G, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Inadequate weight gain in overweight and obese pregnant women: what is the effect on fetal growth? Am J Obstet Gynecol. 2014 Aug;211(2):137.e1-7. doi: 10.1016/j.ajog.2014.02.004. Epub 2014 Feb 11. PMID 24530820
- [Background] Wallace JM, Bhattacharya S, Campbell DM, Horgan GW. Inter-pregnancy weight change impacts placental weight and is associated with the risk of adverse pregnancy outcomes in the second pregnancy. BMC Pregnancy Childbirth. 2014 Jan 22;14:40. doi: 10.1186/1471-2393-14-40. PMID 24450357
- [Background] Jain AP, Gavard JA, Rice JJ, Catanzaro RB, Artal R, Hopkins SA. The impact of interpregnancy weight change on birthweight in obese women. Am J Obstet Gynecol. 2013 Mar;208(3):205.e1-7. doi: 10.1016/j.ajog.2012.12.018. Epub 2012 Dec 12. PMID 23246318
- [Background] Ehrlich SF, Hedderson MM, Feng J, Davenport ER, Gunderson EP, Ferrara A. Change in body mass index between pregnancies and the risk of gestational diabetes in a second pregnancy. Obstet Gynecol. 2011 Jun;117(6):1323-1330. doi: 10.1097/AOG.0b013e31821aa358. PMID 21606742
- [Background] Mostello D, Jen Chang J, Allen J, Luehr L, Shyken J, Leet T. Recurrent preeclampsia: the effect of weight change between pregnancies. Obstet Gynecol. 2010 Sep;116(3):667-672. doi: 10.1097/AOG.0b013e3181ed74ea. PMID 20733450
- [Background] Getahun D, Ananth CV, Oyelese Y, Chavez MR, Kirby RS, Smulian JC. Primary preeclampsia in the second pregnancy: effects of changes in prepregnancy body mass index between pregnancies. Obstet Gynecol. 2007 Dec;110(6):1319-25. doi: 10.1097/01.AOG.0000292090.40351.30. PMID 18055727
- [Background] Bogaerts A, Van den Bergh BRH, Ameye L, Witters I, Martens E, Timmerman D, Devlieger R. Interpregnancy weight change and risk for adverse perinatal outcome. Obstet Gynecol. 2013 Nov;122(5):999-1009. doi: 10.1097/AOG.0b013e3182a7f63e. PMID 24104777
- [Background] Glazer NL, Hendrickson AF, Schellenbaum GD, Mueller BA. Weight change and the risk of gestational diabetes in obese women. Epidemiology. 2004 Nov;15(6):733-7. doi: 10.1097/01.ede.0000142151.16880.03. PMID 15475723
- [Background] Lovelady CA, Garner KE, Moreno KL, Williams JP. The effect of weight loss in overweight, lactating women on the growth of their infants. N Engl J Med. 2000 Feb 17;342(7):449-53. doi: 10.1056/NEJM200002173420701. PMID 10675424
- [Background] Colleran HL, Lovelady CA. Use of MyPyramid Menu Planner for Moms in a weight-loss intervention during lactation. J Acad Nutr Diet. 2012 Apr;112(4):553-8. doi: 10.1016/j.jand.2011.12.004. PMID 22709705
- [Background] Stendell-Hollis NR, Thompson PA, West JL, Wertheim BC, Thomson CA. A comparison of Mediterranean-style and MyPyramid diets on weight loss and inflammatory biomarkers in postpartum breastfeeding women. J Womens Health (Larchmt). 2013 Jan;22(1):48-57. doi: 10.1089/jwh.2012.3707. Epub 2012 Dec 31. PMID 23276189
- [Background] O'Toole ML, Sawicki MA, Artal R. Structured diet and physical activity prevent postpartum weight retention. J Womens Health (Larchmt). 2003 Dec;12(10):991-8. doi: 10.1089/154099903322643910. PMID 14709187
- [Background] Nascimento SL, Pudwell J, Surita FG, Adamo KB, Smith GN. The effect of physical exercise strategies on weight loss in postpartum women: a systematic review and meta-analysis. Int J Obes (Lond). 2014 May;38(5):626-35. doi: 10.1038/ijo.2013.183. Epub 2013 Sep 19. PMID 24048142
- [Background] Rono K, Stach-Lempinen B, Klemetti MM, Kaaja RJ, Poyhonen-Alho M, Eriksson JG, Koivusalo SB; RADIEL group. Prevention of gestational diabetes through lifestyle intervention: study design and methods of a Finnish randomized controlled multicenter trial (RADIEL). BMC Pregnancy Childbirth. 2014 Feb 14;14:70. doi: 10.1186/1471-2393-14-70. PMID 24524674
- [Background] Villamor E, Cnattingius S. Interpregnancy weight change and risk of adverse pregnancy outcomes: a population-based study. Lancet. 2006 Sep 30;368(9542):1164-70. doi: 10.1016/S0140-6736(06)69473-7. PMID 17011943
- [Background] Lassance L, Haghiac M, Leahy P, Basu S, Minium J, Zhou J, Reider M, Catalano PM, Hauguel-de Mouzon S. Identification of early transcriptome signatures in placenta exposed to insulin and obesity. Am J Obstet Gynecol. 2015 May;212(5):647.e1-11. doi: 10.1016/j.ajog.2015.02.026. Epub 2015 Feb 28. PMID 25731694
- [Background] Yassine HN, Marchetti CM, Krishnan RK, Vrobel TR, Gonzalez F, Kirwan JP. Effects of exercise and caloric restriction on insulin resistance and cardiometabolic risk factors in older obese adults--a randomized clinical trial. J Gerontol A Biol Sci Med Sci. 2009 Jan;64(1):90-5. doi: 10.1093/gerona/gln032. Epub 2009 Jan 20. PMID 19164269
- [Background] Institute of Medicine (US) and National Research Council (US) Committee to Reexamine IOM Pregnancy Weight Guidelines; Rasmussen KM, Yaktine AL, editors. Weight Gain During Pregnancy: Reexamining the Guidelines. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32813/ PMID 20669500
- [Background] Resi V, Basu S, Haghiac M, Presley L, Minium J, Kaufman B, Bernard S, Catalano P, Hauguel-de Mouzon S. Molecular inflammation and adipose tissue matrix remodeling precede physiological adaptations to pregnancy. Am J Physiol Endocrinol Metab. 2012 Oct 1;303(7):E832-40. doi: 10.1152/ajpendo.00002.2012. Epub 2012 Jul 17. PMID 22811467
- [Background] Catalano PM, Tyzbir ED, Roman NM, Amini SB, Sims EA. Longitudinal changes in insulin release and insulin resistance in nonobese pregnant women. Am J Obstet Gynecol. 1991 Dec;165(6 Pt 1):1667-72. doi: 10.1016/0002-9378(91)90012-g. PMID 1750458
- [Background] Catalano PM, Tyzbir ED, Wolfe RR, Roman NM, Amini SB, Sims EA. Longitudinal changes in basal hepatic glucose production and suppression during insulin infusion in normal pregnant women. Am J Obstet Gynecol. 1992 Oct;167(4 Pt 1):913-9. doi: 10.1016/s0002-9378(12)80011-1. PMID 1415425
- [Background] Catalano PM, Tyzbir ED, Wolfe RR, Calles J, Roman NM, Amini SB, Sims EA. Carbohydrate metabolism during pregnancy in control subjects and women with gestational diabetes. Am J Physiol. 1993 Jan;264(1 Pt 1):E60-7. doi: 10.1152/ajpendo.1993.264.1.E60. PMID 8430789
- [Background] Catalano PM, Drago NM, Amini SB. Factors affecting fetal growth and body composition. Am J Obstet Gynecol. 1995 May;172(5):1459-63. doi: 10.1016/0002-9378(95)90478-6. PMID 7755054
- [Background] Catalano PM, Drago NM, Amini SB. Maternal carbohydrate metabolism and its relationship to fetal growth and body composition. Am J Obstet Gynecol. 1995 May;172(5):1464-70. doi: 10.1016/0002-9378(95)90479-4. PMID 7755055
- [Background] Catalano PM, Roman-Drago NM, Amini SB, Sims EA. Longitudinal changes in body composition and energy balance in lean women with normal and abnormal glucose tolerance during pregnancy. Am J Obstet Gynecol. 1998 Jul;179(1):156-65. doi: 10.1016/s0002-9378(98)70267-4. PMID 9704782
- [Background] Catalano PM, Huston L, Amini SB, Kalhan SC. Longitudinal changes in glucose metabolism during pregnancy in obese women with normal glucose tolerance and gestational diabetes mellitus. Am J Obstet Gynecol. 1999 Apr;180(4):903-16. doi: 10.1016/s0002-9378(99)70662-9. PMID 10203659
- [Background] Catalano PM, Nizielski SE, Shao J, Preston L, Qiao L, Friedman JE. Downregulated IRS-1 and PPARgamma in obese women with gestational diabetes: relationship to FFA during pregnancy. Am J Physiol Endocrinol Metab. 2002 Mar;282(3):E522-33. doi: 10.1152/ajpendo.00124.2001. PMID 11832353
- [Background] O'Tierney-Ginn P, Presley L, Myers S, Catalano P. Placental growth response to maternal insulin in early pregnancy. J Clin Endocrinol Metab. 2015 Jan;100(1):159-65. doi: 10.1210/jc.2014-3281. PMID 25365315
- [Background] Koontz MB, Gunzler DD, Presley L, Catalano PM. Longitudinal changes in infant body composition: association with childhood obesity. Pediatr Obes. 2014 Dec;9(6):e141-4. doi: 10.1111/ijpo.253. Epub 2014 Sep 30. PMID 25267097
- [Background] Kirwan JP, Varastehpour A, Jing M, Presley L, Shao J, Friedman JE, Catalano PM. Reversal of insulin resistance postpartum is linked to enhanced skeletal muscle insulin signaling. J Clin Endocrinol Metab. 2004 Sep;89(9):4678-84. doi: 10.1210/jc.2004-0749. PMID 15356080
- [Background] Friedman JE, Kirwan JP, Jing M, Presley L, Catalano PM. Increased skeletal muscle tumor necrosis factor-alpha and impaired insulin signaling persist in obese women with gestational diabetes mellitus 1 year postpartum. Diabetes. 2008 Mar;57(3):606-13. doi: 10.2337/db07-1356. Epub 2007 Dec 14. PMID 18083784
- [Background] Solomon TP, Haus JM, Kelly KR, Rocco M, Kashyap SR, Kirwan JP. Improved pancreatic beta-cell function in type 2 diabetic patients after lifestyle-induced weight loss is related to glucose-dependent insulinotropic polypeptide. Diabetes Care. 2010 Jul;33(7):1561-6. doi: 10.2337/dc09-2021. Epub 2010 Mar 3. PMID 20200305
- [Background] Solomon TP, Haus JM, Kelly KR, Cook MD, Filion J, Rocco M, Kashyap SR, Watanabe RM, Barkoukis H, Kirwan JP. A low-glycemic index diet combined with exercise reduces insulin resistance, postprandial hyperinsulinemia, and glucose-dependent insulinotropic polypeptide responses in obese, prediabetic humans. Am J Clin Nutr. 2010 Dec;92(6):1359-68. doi: 10.3945/ajcn.2010.29771. Epub 2010 Oct 27. PMID 20980494
- [Background] Calabuig-Navarro V, Puchowicz M, Glazebrook P, Haghiac M, Minium J, Catalano P, Hauguel deMouzon S, O'Tierney-Ginn P. Effect of omega-3 supplementation on placental lipid metabolism in overweight and obese women. Am J Clin Nutr. 2016 Apr;103(4):1064-72. doi: 10.3945/ajcn.115.124651. PMID 26961929
- [Background] Ptomey LT, Willis EA, Honas JJ, Mayo MS, Washburn RA, Herrmann SD, Sullivan DK, Donnelly JE. Validity of energy intake estimated by digital photography plus recall in overweight and obese young adults. J Acad Nutr Diet. 2015 Sep;115(9):1392-9. doi: 10.1016/j.jand.2015.05.006. Epub 2015 Jun 26. PMID 26122282
- [Background] Look AHEAD Research Group; Wadden TA, West DS, Delahanty L, Jakicic J, Rejeski J, Williamson D, Berkowitz RI, Kelley DE, Tomchee C, Hill JO, Kumanyika S. The Look AHEAD study: a description of the lifestyle intervention and the evidence supporting it. Obesity (Silver Spring). 2006 May;14(5):737-52. doi: 10.1038/oby.2006.84. PMID 16855180
- [Background] Donnelly JE, Goetz J, Gibson C, Sullivan DK, Lee R, Smith BK, Lambourne K, Mayo MS, Hunt S, Lee JH, Honas JJ, Washburn RA. Equivalent weight loss for weight management programs delivered by phone and clinic. Obesity (Silver Spring). 2013 Oct;21(10):1951-9. doi: 10.1002/oby.20334. Epub 2013 May 25. PMID 23408579
- [Background] Siri WE. Body composition from fluid spaces and density: analysis of methods. 1961. Nutrition. 1993 Sep-Oct;9(5):480-91; discussion 480, 492. No abstract available. PMID 8286893
- [Background] Catalano PM, Wong WW, Drago NM, Amini SB. Estimating body composition in late gestation: a new hydration constant for body density and total body water. Am J Physiol. 1995 Jan;268(1 Pt 1):E153-8. doi: 10.1152/ajpendo.1995.268.1.E153. PMID 7840173
- [Background] Sady SP, Carpenter MW, Sady MA, Haydon B, Hoegsberg B, Cullinane EM, Thompson PD, Coustan DR. Prediction of VO2max during cycle exercise in pregnant women. J Appl Physiol (1985). 1988 Aug;65(2):657-61. doi: 10.1152/jappl.1988.65.2.657. PMID 3170418
- [Background] Watanabe RM, Steil GM, Bergman RN. Critical evaluation of the combined model approach for estimation of prehepatic insulin secretion. Am J Physiol. 1998 Jan;274(1):E172-83. doi: 10.1152/ajpendo.1998.274.1.E172. PMID 9458763
- [Background] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898
- [Background] Jacobson AM, de Groot M, Samson JA. The evaluation of two measures of quality of life in patients with type I and type II diabetes. Diabetes Care. 1994 Apr;17(4):267-74. doi: 10.2337/diacare.17.4.267. PMID 8026281
- [Background] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- [Background] Sewell MF, Huston-Presley L, Super DM, Catalano P. Increased neonatal fat mass, not lean body mass, is associated with maternal obesity. Am J Obstet Gynecol. 2006 Oct;195(4):1100-3. doi: 10.1016/j.ajog.2006.06.014. Epub 2006 Jul 26. PMID 16875645
- [Background] Catalano PM, Tyzbir ED, Allen SR, McBean JH, McAuliffe TL. Evaluation of fetal growth by estimation of neonatal body composition. Obstet Gynecol. 1992 Jan;79(1):46-50. PMID 1727584
- [Background] Catalano PM, Thomas AJ, Avallone DA, Amini SB. Anthropometric estimation of neonatal body composition. Am J Obstet Gynecol. 1995 Oct;173(4):1176-81. doi: 10.1016/0002-9378(95)91348-3. PMID 7485315
- [Background] Catalano PM, Presley L, Minium J, Hauguel-de Mouzon S. Fetuses of obese mothers develop insulin resistance in utero. Diabetes Care. 2009 Jun;32(6):1076-80. doi: 10.2337/dc08-2077. PMID 19460915
- [Background] Lindsay CA, Thomas AJ, Catalano PM. The effect of smoking tobacco on neonatal body composition. Am J Obstet Gynecol. 1997 Nov;177(5):1124-8. doi: 10.1016/s0002-9378(97)70027-9. PMID 9396906
- [Background] Rohl J, Huston-Presley L, Amini S, Stepanchak B, Catalano P. Factors associated with fetal growth and body composition as measured by ultrasound. Am J Obstet Gynecol. 2001 Dec;185(6):1416-20. doi: 10.1067/mob.2001.118846. PMID 11744918
- [Background] Hashimoto K, Wong WW, Thomas AJ, Uvena-Celebrezze J, Huston-Pressley L, Amini SB, Catalano PM. Estimation of neonatal body composition: isotope dilution versus total-body electrical conductivity. Biol Neonate. 2002;81(3):170-5. doi: 10.1159/000051530. PMID 11937722
- [Background] Uvena-Celebrezze J, Fung C, Thomas AJ, Hoty A, Huston-Presley L, Amini SB, Catalano PM. Relationship of neonatal body composition to maternal glucose control in women with gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2002 Dec;12(6):396-401. doi: 10.1080/jmf.12.6.396.401. PMID 12683650
- [Background] Catalano PM, Thomas A, Huston-Presley L, Amini SB. Increased fetal adiposity: a very sensitive marker of abnormal in utero development. Am J Obstet Gynecol. 2003 Dec;189(6):1698-704. doi: 10.1016/s0002-9378(03)00828-7. PMID 14710101
- [Background] Durnwald C, Huston-Presley L, Amini S, Catalano P. Evaluation of body composition of large-for-gestational-age infants of women with gestational diabetes mellitus compared with women with normal glucose tolerance levels. Am J Obstet Gynecol. 2004 Sep;191(3):804-8. doi: 10.1016/j.ajog.2003.11.033. PMID 15467545
- [Background] Singh KA, Huston-Presley LP, Mencin P, Thomas A, Amini SB, Catalano PM. Birth weight and body composition of neonates born to Caucasian compared with African-American mothers. Obstet Gynecol. 2010 May;115(5):998-1002. doi: 10.1097/AOG.0b013e3181da901a. PMID 20410774
- [Background] Waters TP, Huston-Presley L, Catalano PM. Neonatal body composition according to the revised institute of medicine recommendations for maternal weight gain. J Clin Endocrinol Metab. 2012 Oct;97(10):3648-54. doi: 10.1210/jc.2012-1781. Epub 2012 Jul 20. PMID 22821895
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Lassance L, Haghiac M, Minium J, Catalano P, Hauguel-de Mouzon S. Obesity-induced down-regulation of the mitochondrial translocator protein (TSPO) impairs placental steroid production. J Clin Endocrinol Metab. 2015 Jan;100(1):E11-8. doi: 10.1210/jc.2014-2792. PMID 25322273
- [Background] Visiedo F, Bugatto F, Sanchez V, Cozar-Castellano I, Bartha JL, Perdomo G. High glucose levels reduce fatty acid oxidation and increase triglyceride accumulation in human placenta. Am J Physiol Endocrinol Metab. 2013 Jul 15;305(2):E205-12. doi: 10.1152/ajpendo.00032.2013. Epub 2013 May 14. PMID 23673156
- [Background] Brass E, Hanson E, O'Tierney-Ginn PF. Placental oleic acid uptake is lower in male offspring of obese women. Placenta. 2013 Jun;34(6):503-9. doi: 10.1016/j.placenta.2013.03.009. Epub 2013 Apr 17. PMID 23602336
- [Background] Hughes SD, Quaade C, Johnson JH, Ferber S, Newgard CB. Transfection of AtT-20ins cells with GLUT-2 but not GLUT-1 confers glucose-stimulated insulin secretion. Relationship to glucose metabolism. J Biol Chem. 1993 Jul 15;268(20):15205-12. PMID 8325893
- [Background] FOLCH J, LEES M, SLOANE STANLEY GH. A simple method for the isolation and purification of total lipides from animal tissues. J Biol Chem. 1957 May;226(1):497-509. No abstract available. PMID 13428781
- [Background] Erickson ML, Mey JT, Axelrod CL, Paul D, Gordesky L, Russell K, Barkoukis H, O'Tierney-Ginn P, Fielding RA, Kirwan JP, Catalano PM. Rationale and study design for lifestyle intervention in preparation for pregnancy (LIPP): A randomized controlled trial. Contemp Clin Trials. 2020 Jul;94:106024. doi: 10.1016/j.cct.2020.106024. Epub 2020 May 8. PMID 32389808

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT03146156/Prot_SAP_000.pdf